CLINICAL TRIAL: NCT06271863
Title: Outcome of Conservative Management in Cases of Pre Mature Rupture of Membranes (PROM) Between 20 and 28 Weeks of Pregnancy in Sohag City Hospitals
Status: Enrolling by invitation | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mahmoud Nabil Halabi, Resident, Sohag University
Other Study IDs: Soh-Med-23-11-08MS
Record Dates: First submitted 2024-02-06; First posted 2024-02-22 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: PROM, Preterm (Pregnancy)
MeSH Terms: conditions — Fetal Membranes, Premature Rupture

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — CBC , CRP ,
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Prospective observational study

ELIGIBILITY:
Inclusion Criteria:

* pregnant woman 24 weeks to 28 weeks of pregnancy with PROM

Exclusion Criteria:

* gestational age other than the mentioned before Multiple pregnancy Cerclage Other causes of decreased AF

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: pregnant woman 24 weeks to 28 weeks of pregnancy with PROM in sohag city hospitals
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Conservation vs termination in cases of PROM 20 to 28 weeks of pregnancy | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided